CLINICAL TRIAL: NCT01111474
Title: Effectiveness of Cyanoacrylate and Laser in the Treatment of Cervical Dentin Sensitivity
Brief Title: Cyanoacrylate and Laser and Dentin Sensitivity
Acronym: Cyano-laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Principal Investigator, Olga Flecha, PHD student, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: odf2008
Record Dates: First submitted 2010-04-20; First posted 2010-04-27 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Dentin Hypersensitivity; Dentin Sensitivity
Keywords: dentin hypersensitivity; cyanoacrylate; laser
MeSH Terms: conditions — Dentin Sensitivity | interventions — Cyanoacrylates; Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyanoacrylate (Active Comparator): 3 applications of cyanoacrylate (48 hours interval)at the cervical region of the sensitive tooth
  Interventions: Other: Cyanoacrylate
- Laser (Active Comparator): 3 Low intensity laser application (48 hour interval). The application of 1Joule/cm^2 was performed for eight seconds at three points along the dental neck, using the infrared wavelength (795nm)
  Interventions: Radiation: Laser

INTERVENTIONS:
Other: Cyanoacrylate — 3 applications of cyanoacrylate (48 hours interval) at the cervical region of the sensitive tooth
  Other Names: Superbonder
  Arms: Cyanoacrylate
Radiation: Laser — This process was conducted three times with an interval of 48 hours between applications, according to laser's manufacturer advice Clean Line Easy Laser - LILT®, Clean Line Easy Laser Doctor Dental Products Industry LTDA, BRA). For dentin hypersensitivity, the application of 1Joule/cm^2 is recommended for eight seconds at three points along the dental neck, using the infrared wavelength (795nm).
  Other Names: LILT
  Arms: Laser

SUMMARY:
This study aimed to evaluate the effectiveness of two treatments for dental hypersensitivity: cyanoacrylate (Super Bonder®) compared with use of low intensity laser treatment (LILT). As the cyanoacrylate is a lower cost treatment, the hypothesis in investigation is if this product is equally effective as the laser treatment.

DETAILED DESCRIPTION:
The present study included 62 patients (15 male and 47 females, aged 12 to 60 years). The initial cervical dentin hypersensitivity was checked throughout a thermal test (air blast). The 434 teeth included were that with a score ≥5 in a numerical scale rating of pain. Teeth were randomly assigned according quadrants (split mouth design) - 216 were allocated to LILT group and 218 for the Super Bonder® group. Thermal tests with a tetrafluoroethane spray (Endo-Ice®) and air blast were performed and considered as baseline. Pain parameters were recorded using a numerical scale rating with 24 hours, 30, 90 and 180 days after the interventions. Quality of life of the patients was also assessed with the use of OHIP-14 at baseline and after 180 days.

ELIGIBILITY:
Inclusion Criteria:

1. patients should be in good general and dental health;
2. present complaints of dental sensitivity to cold, sweet, acidic foods and brushing;
3. present complaints of pain in teeth located in different quadrants;
4. manifest pain or discomfort upon application of the triple syringe air jet;
5. not be in current use of desensitizing agents.

Exclusion Criteria:

1. presence of extensive restorations and carious lesions in the sensitive teeth;
2. undergoing orthodontic treatment;
3. frequent use of analgesics, antidepressants and anti-inflammatory drugs;
4. presence of gingival inflammation;
5. non-consent of patient.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga D. Flecha, pHD student, Principal Investigator — UNIFESP - Federal University of São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients with dentin hypersensitivity were recruited through posters and folders provided at the Dental Clinics, schools, gyms and drugstores.
Pre-assignment Details: The patients which had not achieved an initial level of hypersensitivity were excluded from the trial before assignment to the groups.
Groups:
- All Study Participants: In this split mouth study, teeth from the participants were randomly assigned according to quadrants, to either receive Cyanoacrilate (Superbonder) or Laser (LILT). Cyanoacrylate: 3 applications with a microbrush (48 hour interval). Laser: 3 Low intensity laser application (48 hour interval). The application of 1Joules/cm^2 was performed for eight seconds at three points along the dental neck, using the infrared wavelength (795nm)
Period: Overall Study
Arm/Group | All Study Participants
Started | 74 (593 teeth from 74 participants: 296 teeth treated with cyanoacrylate and 297 teeth with LILT)
Completed | 62 (434 teeth from 62 participants: 218 teeth teated with cyanoacrylate and 216 teeth with LILT)
Not Completed | 12
Not completed — Lost to Follow-up | 12

BASELINE CHARACTERISTICS:
Population: 62 participants contributed with 434 teeth in a split mouth design: 216 teeth were treated with laser and 218 teeth were treated with cyanoacrylate.
Groups:
- All Study Participants: In this split mouth study, teeth from the participants were randomly assigned according to quadrants, to either receive Cyanoacrylate (Superbonder) or Laser (LILT).
  Cyanoacrylate: 3 applications of Superbonder (48 hours interval) at the cervical region of the sensitive tooth. LILT: 3 Low intensity laser application (48 hour interval). The application of 1Joules/cm^2 was performed for eight seconds at three points along the dental neck, using the infrared wavelength (795nm)
Arm/Group | All Study Participants
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (10.7)
Sex/Gender, Customized [Number; unit: participants]
  Male | 15
  Female | 47

OUTCOME MEASURES:

1. Primary Outcome: Change of the Pain Sensitivity
Description: Change in pain experienced by the participants was calculated as the difference between baseline level of pain sensitivity and after 180 days. Pain was recorded using a numerical pain assessment scale with range between 0 (no pain) to 10 (worst possible pain). The higher the numbering the worse the result.
Time Frame: Baseline and 180 days
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: teeth
Arm/Group | Cyanoacrylate | Laser
Number analyzed (Participants) | 62 | 62
Number analyzed (teeth) | 218 | 216
score on a scale
  Baseline | 7.77 (1.7) | 7.49 (1.7)
  180 days | 2.57 (2.9) | 2.36 (2.7)

2. Secondary Outcome: Quality of Life Improvement
Description: Difference between the level of quality of life - Oral Health Impact Profile "OHIP" at baseline and 180 days. OHIP-14 total scale ranges from 0 to 56 points with higher scores indicating a poorer oral health-related quality of life. The response format uses a Likert-type frequency scale such as follows: very often = 4, fairly often = 3, occasionally = 2, hardly ever = 1, never = 0. Total score is obtained by summing the response codes of the 14 items constituting the measure.
Time Frame: Baseline and 180 days
Population: 62 participants contributed with 62 questionnaires in each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cyanoacrylate | Laser
Number analyzed (Participants) | 62 | 62
score on a scale
  Baseline | 16.87 (9.1) | 16.87 (9.1)
  180 days | 12.05 (8.0) | 12.05 (8.0)

ADVERSE EVENTS:
Groups:
- Laser: 3 Low intensity laser application (48 hour interval). The application of 1J/cm2 was performed for eight seconds at three points along the dental neck, using the infrared wavelength (660nm)
Arm/Group | Cyanoacrylate | Laser
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No